CLINICAL TRIAL: NCT03630367
Title: Effects of Adding L-Carnitine With Dexamethasone on Respiratory Distress Syndrome Development in Preterm Infants
Brief Title: Effects of L-Carnitine Supplementation on Respiratory Distress Syndrome
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Unavailability of the medication
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LCPET
Record Dates: First submitted 2018-08-04; First posted 2018-08-14 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Premature Birth
MeSH Terms: conditions — Premature Birth | interventions — Dexamethasone; Carnitine; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): women will receive dexamethasone 8 mg intramuscular every 8 hours plus single injection of L-carnitine 1 gm slow intravenous
  Interventions: Drug: Dexamethasone; Drug: L-Carnitine 1G/5mL Injection
- control group (Active Comparator): women will receive dexamethasone 8 mg intramuscular every 8 hours plus single injection of saline 1 gm slow intravenous
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Intramuscular injection 8 mg
Drug: L-Carnitine 1G/5mL Injection — slow intravenous injection
  Arms: study group

SUMMARY:
The aim of the present study was to investigate the efficacy of L-carnitine therapy on the occurrence and prognosis of respiratory distress syndrome

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 30-37 weeks
* singleton pregnancy

Exclusion Criteria:

* congenital malformed fetus
* Extreme premature

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
the mean difference in the Apgar score after birth | 1 minute
  Assessment of fetal general condition

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt